CLINICAL TRIAL: NCT03577808
Title: Validation of Organoids Potential Use as a Companion Diagnostic in Predicting Neoadjuvant Chemoradiation Sensitivity in Locally Advanced Rectal Cancer
Brief Title: Organoids in Predicting Chemoradiation Sensitivity on Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhen Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhen Zhang, Professor Zhang, Fudan University
Organization: Fudan University (Other)
Other Study IDs: FDRT-R008
Record Dates: First submitted 2018-06-20; First posted 2018-07-05 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Organoids; Rectal Cancer; Chemoradiation
MeSH Terms: conditions — Rectal Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arm: Patients with locally advanced rectal cancer will receive neoadjuvant chemoradiation. The radiation procedure and concurrent chemotherapy drugs will base on clinical practice. Organoids bio-bank of pre-treatment tumor biopsies will be established and exposed to irradiation and the same chemotherapy drugs as the corresponding patient.
  Interventions: Other: Biopsy

INTERVENTIONS:
Other: Biopsy — Patients with locally advanced rectal cancer will receive biopsy of the primary tumor before neoadjuvant chemoradiation.

SUMMARY:
Patients with locally advanced rectal cancer will receive biopsy before the standard treatment of neoadjuvant chemoradiation. The investigators are going to establish organoids model from the pre-treatment biopsies and expose organoids to irradiation and the same chemotherapy drugs. The sensitivity of irradiation and chemotherapy drugs will be tested in the organoids model. Here, the investigators will launch the observational clinical trial to validate whether the organoids could predict the clinical outcome in locally advanced rectal cancer patients underwent neoadjuvant chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

* pathological confirmed adenocarcinoma
* clinical stage T3-4 and/or N+
* the distance from anal verge less than 12 cm
* without distance metastases
* KPS >=70
* without previous anti-cancer therapy
* sign the inform consent

Exclusion Criteria:

* pregnancy or breast-feeding women
* serious medical illness
* baseline blood and biochemical indicators do not meet the following criteria: neutrophils≥1.5×10^9/L, Hb≥90g/L, PLT≥100×10^9/L, ALT/AST ≤2.5 ULN, Cr≤ 1 ULN

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced rectal cancer will receive neoadjuvant chemoradiation. The radiation procedure and concurrent chemotherapy drugs will base on clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-08-17 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Response of the rectal cancer organoids to irradiation and the same chemotherapy drugs as the corresponding patient. | 2018.08-2020.11
  The investigators will culture rectal cancer organoids and treat with irradiation and the same chemotherapy drugs as the corresponding patient. The number and size of alive organoids will be observed after treatment. The correlation of organoids sensitivity and patient response will be evaluated.

SECONDARY OUTCOMES:
Response of the rectal cancer patients to neoadjuvant chemoradiation. | 2018.08-2020.11
  The investigators will use pathological tumor regression grade (TRG) to evaluate chemoradiation response of locally advanced rectal cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, MD, Principal Investigator — Fudan University; Guoqiang Hua, PhD, Principal Investigator — Institute of Radiation Medicine, Fudan University
Locations (1):
- Fudan University, Shanghai, China